CLINICAL TRIAL: NCT06489509
Title: Distribution of Pulmonary Ventilation in Lateral Decubitus of Healthy Adults Under Non-Invasive Mechanical Ventilation Supply
Brief Title: Distribution of Pulmonary Ventilation in Lateral Decubitus of Healthy Adults Under Non-Invasive Mechanical Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Konstantinos Grigoriadis, Chief of allied health professions, Attikon Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: EBD2878
Record Dates: First submitted 2024-06-26; First posted 2024-07-08 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Noninvasive Ventilation; Patient Positioning
Keywords: impedance tomography; distribution of ventilation; lateral decubitus; Noninvasive Ventilation

STUDY DESIGN:
Intervention Model Description: The regional distribution of pulmonary ventilation was measured in the supine, right, and left lateral positions while alternating the sides to ensure randomization.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Supine position (Active Comparator): Supine experimental position
  Interventions: Device: Positive End Expiratory Pressure 5 H2O; Device: Positive End Expiratory Pressure 10 H2O
- Right position (Active Comparator): Right lateral decubitus
  Interventions: Device: Positive End Expiratory Pressure 5 H2O; Device: Positive End Expiratory Pressure 10 H2O
- Left position (Active Comparator): Left lateral decubitus
  Interventions: Device: Positive End Expiratory Pressure 5 H2O; Device: Positive End Expiratory Pressure 10 H2O

INTERVENTIONS:
Device: Positive End Expiratory Pressure 5 H2O — Positive End Expiratory Pressure 5 H2O from CPAP apparatus
Device: Positive End Expiratory Pressure 10 H2O — Positive End Expiratory Pressure 5 H2O from CPAP apparatus

SUMMARY:
The aim was to investigate via impedance tomography apparatus the distribution of pulmonary ventilation at a lateral position at different Continuous Positive Airway Pressure levels (0, 5, 10 cm Η2Ο) in healthy subjects.

DETAILED DESCRIPTION:
In lateral decubitus, the largest percentage of pulmonary ventilation of non-sedated subjects is distributed mainly in the dependent lung. The aim It was to investigate via impedance tomography apparatus the distribution of pulmonary ventilation at a lateral position at different Continuous Positive Airway Pressure levels (0, 5, 10 cm Η2Ο) in healthy subjects. The volunteers were noninvasively ventilated in both lateral positions and supine positions at the beginning and end of the process. It is concluded that implementing Non-Invasive Ventilation in the lateral body position resulted in increased ventilation of the dependent lung. In contrast, the respective ventilation of the non-dependent lung was further decreased.

ELIGIBILITY:
Inclusion Criteria:

• Healthy Volunteers

Exclusion Criteria:

* Chronic respiratory disease
* BMI>40
* Smoking history

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2018-07-08 (Actual); Study Completion 2018-07-08 (Actual)

PRIMARY OUTCOMES:
The percentage change in pulmonary ventilation | Up to 3 minutes
  The percentage change in pulmonary ventilation was measured at each position, without applying external positive end-expiratory pressure and under positive end-expiratory pressure of 5 and 10 cmH2O

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Grigoriadis, Dr, Principal Investigator — PT, Attikon University Hospital; Anna Grigoriadou, MSc, Study Director — PT, Attikon University Hospital; Frantzeska Frantzeskaki, Study Director — MD, Attikon University Hospital; Ioannis Efstathiou, Study Director — PT, Attikon University Hospital; Iraklis Tsangaris, Study Chair — Professor, Attikon University Hospital
Locations (2):
- Greece (2):
  - Attikon University Hospital, Athens, Attica
  - Grigoriadis Konstantinos, Athens, Attica

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schnidrig S, Casaulta C, Schibler A, Riedel T. Influence of end-expiratory level and tidal volume on gravitational ventilation distribution during tidal breathing in healthy adults. Eur J Appl Physiol. 2013 Mar;113(3):591-8. doi: 10.1007/s00421-012-2469-7. Epub 2012 Aug 8. PMID 22872368
- [Background] Sharma JP, Salhotra R, Kumar S, Tyagi A, Sethi AK. Noninvasive lung recruitment maneuver prevents reintubation and reduces ICU stay. Lung India. 2016 Jan-Feb;33(1):99-101. doi: 10.4103/0970-2113.173070. No abstract available. PMID 26933321
- [Result] Hurewitz AN, Susskind H, Harold WH. Obesity alters regional ventilation in lateral decubitus position. J Appl Physiol (1985). 1985 Sep;59(3):774-83. doi: 10.1152/jappl.1985.59.3.774. PMID 4055566
- [Result] Lobo B, Hermosa C, Abella A, Gordo F. Electrical impedance tomography. Ann Transl Med. 2018 Jan;6(2):26. doi: 10.21037/atm.2017.12.06. PMID 29430443
- [Result] Miura MC, Ribeiro de Carvalho CR, Yamada da Silveira LT, de Moraes Regenga M, Petri Damiani L, Fu C. The effects of recruitment maneuver during noninvasive ventilation after coronary bypass grafting: A randomized trial. J Thorac Cardiovasc Surg. 2018 Dec;156(6):2170-2177.e1. doi: 10.1016/j.jtcvs.2018.05.004. Epub 2018 May 28. PMID 29945735
- [Result] Nishimura M. Electrical Impedance Tomography: The Promise of Noninvasive Lung Images at the Bedside. Respir Care. 2020 Mar;65(3):402-403. doi: 10.4187/respcare.07716. No abstract available. PMID 32086337